CLINICAL TRIAL: NCT05159024
Title: A Prospective Cohort Study on the Role of The Triad of Procalcitonin, C-Reactive Protein, and White Blood Cell Count in The Prediction of Anastomotic Leak Following Colorectal Resections
Brief Title: Role of Procalcitonin, C-Reactive Protein, and WBC Count in Prediction of Colorectal Anastomotic Leak
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Waleed Ghareeb, Lecturer of surgery, Suez Canal University
Other Study IDs: Trajectory2021
Record Dates: First submitted 2021-11-18; First posted 2021-12-15 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with leak after colorectal anastomosis: Patients who developed anastomotic leak, clinical or radiologic, after colorectal resection and anastomosis
  Interventions: Diagnostic Test: CRP, PCT, and WBCs trajectories

INTERVENTIONS:
Diagnostic Test: CRP, PCT, and WBCs trajectories — the levels of CRP, PCT, and WBCs were assessed before surgery and after the onset of leak

SUMMARY:
The interest in identifying a biological marker for the early detection of AL is growing. Such a marker could play a vital role in modern fast-track multimodal protocols, allowing safe and early discharge of patients after colorectal surgery with a low rate of readmission. C-reactive protein (CRP) has been identified as a valid parameter for detection of postoperative infectious complications after rectal resection. A serum CRP level greater than 12.4 mg/dL on postoperative day (POD) 4 is considered predictive of septic complications. According to a recent analysis, the changes in the trajectory of CRP levels might be more beneficial than a snipped point. Moreover, the trajectory has a negative predictability of up to 99.3%. Another interesting biomarker is procalcitonin (PCT), the prohormone of calcitonin, produced by parafollicular C cells in the thyroid. Normally, it has a very low plasma concentration in healthy individuals (0.01-0.05 ng/mL), and it increases during severe generalized bacterial, parasitic, or fungal infections, but not in noninfectious inflammatory reactions. Procalcitonin has been described as an early, sensitive, and specific marker of sepsis. Moreover, the plasma concentration of PCT has been used as an early predictor of infection in acute pancreatitis, secondary peritonitis, and infectious complications after thoracic, esophageal, and cardiac surgeries. In addition, elevated white blood cell (WBC) count is associated with AL after gastrointestinal surgeries. Therefore, this study was conducted to evaluate the utility of CRP, PCT, and WBC count trajectories, as separate and combined biomarkers for prediction of AL after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of either sex who underwent colorectal surgery entailing an anastomosis

Exclusion Criteria:

* Patients younger than 18 years
* Patients with active infection at the time of surgery
* Patients who had received chemotherapy or radiotherapy
* Patients on long-term corticosteroid therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 205 patients who had colorectal surgery, all patients had a diagnosis of new or previous colorectal cancer. 56.1% of patients were males and 43.9% were females. Patient age ranged from 25 to 78 years, with a mean of 56.4 years
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of combined CRP-PCT- WBC trajectory in prediction of anastomotic leak | five days after surgery
  Sensitivity, specificity and accuracy of combined CRP-PCT- WBCs trajectory

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided